CLINICAL TRIAL: NCT06039241
Title: Prospective, Non-interventional, Observational Study for Multi-dimensional Assessment of Signs, Symptoms, Quality of Life and Disease Control of Long-term Treatment With Dupilumab in Patients With Atopic Dermatitis (≥6 Years)
Brief Title: Real-world Effectiveness Study of Long-term Treatment With Dupilumab in Participants ≥6 Years With Atopic Dermatitis
Acronym: PROTYPE2
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17251; U1111-1293-5998 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-08-07; First posted 2023-09-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AD patients treated with dupilumab: Patients ≥6 years of age in whom dupilumab therapy was initiated to treat their severe AD (6-11 years) or moderate to severe AD (adult and adolescent patients ≥12 years of age) based on the patient's medical requirements and standards of best medical practice.

SUMMARY:
This is a Prospective, non-interventional (NIS) observational study in patients (≥6 years) with atopic dermatitis (AD) receiving dupilumab for the prospective evaluation of signs and symptoms, quality of life and disease control. The aim of this NIS is the characterization of the AD patient population in Germany, receiving dupilumab under everyday conditions in terms of their medical history, socio-demographic and disease-related characteristics, associated atopic comorbidities and type 2 inflammation diseases, concomitant therapy as well as previous systemic and ongoing AD treatments. In addition to the therapeutic response rate at Month 6, the long-term efficacy of dupilumab at Month 12 and Month 24 will be assessed by additional outcomes by measuring disease control in AD patients using questionnaires such as Atopic Dermatitis Control Tool (ADCT) and Recap of Atopic Eczema (RECAP). In addition, this NIS aims to assess the dosing pattern of dupilumab for AD, including variations in dosing regimen, reason for dupilumab treatment initiation or discontinuation, or change in therapy and concomitant therapies and duration of treatment. In addition, the effect of dupilumab in adult and pediatric AD patients with associated atopic comorbidities or type-2 inflammation diseases are observed, which corresponds to the clinical care situation. Finally, this NIS aims to collect long-term safety data in adult, adolescent and pediatric AD patients treated with dupilumab. Individual observation period is 2 years or until dupilumab is discontinued. Visits will be scheduled according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients are at least 6 years of age at the baseline visit.
* Initial treatment with dupilumab was initiated in adults and adolescents 12 years of age and older with moderate to severe AD, or in children 6 to 11 years of age with severe AD according to the Summary of Product Characteristics.
* Patients or their guardians are able to understand and complete the study-related questionnaires.
* Signing a written informed consent form by the patients before the initiation of documentation within the framework of this NIS or informed consent of parents/guardian, if applicable.

Exclusion Criteria:

* Patients who have a contraindication for dupilumab based on the current Summary of Product Characteristics.
* Patients who have already been treated with dupilumab for more than 7 days.
* Any acute or chronic diseases, which, in the opinion of the attending physician, would impair the patient's ability to complete questionnaires or participate in this study or could affect the interpretation of the results.
* Participation in an ongoing interventional or observational study, which, in the opinion of the attending physician, could affect the assessment of the current study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥6 years of age in whom dupilumab therapy was initiated to treat their severe AD (6-11 years) or moderate to severe AD (adult and adolescent patients ≥12 years of age) according to the Summary of Product Characteristics. The decision to initiate treatment with dupilumab will be made by the attending physician based on the patient's medical requirements and standards of best medical practice. This decision will be made independent of and prior to data collection in this non-interventional study (NIS).
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-03-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who maintain Eczema Area and Severity Index (EASI) ≤ 7 OR peak pruritus Numerical Rating Scale (NRS) ≤ 4 OR Dermatology Life Quality Index (DLQI) ≤ 5 | From Month 6 to Month 12
  EASI is a Measure used in clinical practice and clinical trials to assess the severity and extent of Atopic Dermatitis (AD). Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity. DLQI is a questionaire with a score system of 0 to 30 the high score is indicative of poor QoL
Mean percent change from baseline in Atopic Dermatitis Control Tools (ADCT) score (≥12 years) | From baseline to Week 52
  Atopic dermatitis control tool (ADCT) is a validated, brief and easy scored tool designed to evaluate patient-perceived control of atopic dermatitis, to foster communication between patients and their physicians and help appropriate decision- making. ADCT questionnaire assess patient-self-perceived control of their AD with a total score from 0 to 24; higher scores indicate lower AD control. ADCT is a questionnaire to assess patient-self-perceived control of their AD with a total score from 0 to 24; higher scores indicate lower AD control.
Mean percent change from baseline in Recap of atopic eczema (RECAP) score (6-11 years) | From baseline to Week 52
  Recap of atopic eczema (RECAP) is a seven-item questionnaire designed to capture the experience of eczema control in all ages and eczema severities. Patient's who turn 12 years during the course of study will continue to complete RECAP.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) during the observation period | From baseline up to 24 months
  Treatment emergent AEs and SAEs reported
Incidence of dupilumab-related TEAEs during the observation period. | From baseline up to 24 months
  Treatment emergent AEs and SAEs reported
Event rate (per patient year) by type of TEAEs during the observation period. | From baseline up to 24 months
Event rate (per patient year) by type of dupilumab related TEAEs during the observational period | From Baseline up to 24 months
Treating physician reported effectiveness data: Change from baseline in IGA score after 6, 12, and 24 months dupilumab therapy | From baseline up to 24 months
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity
Treating physician reported effectiveness data.: Number of patients achieving EASI-75 (improvement in EASI score from baseline of ≥ 75%) after 6, 12 and 24 months of dupilumab therapy | From baseline up to 24 months
  EASI is a Measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders are the participants who achieved ≥75% improvement from baseline.
Treating physician reported effectiveness data: Absolute change from baseline in EASI score after 6, 12 and 24 months of dupilumab therapy | From baseline up to 24 months
  EASI is a Measure used in clinical practice and clinical trials to assess the severity and extent of AD, The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD
Treating physician reported effectiveness data: Percentage change from baseline in EASI score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  EASI is a Measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI score is used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Treating physician reported effectiveness data: Absolute change from baseline in IGA score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Treating physician reported effectiveness data: Change from baseline in body surface area (BSA) after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  Affected body surface area is measured.
Patient reported effectiveness and impact on quality of life (QoL) data: Mean absolute change from baseline in Atopic Dermatitis Control Test (ADCT) score after 3, 6, 9, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  ADCT is a validated, brief and easy scored tool designed to evaluate patient-perceived control of atopic dermatitis, to foster communication between patients and their physicians and help appropriate decision making. The ADCT is a 6-item patient-reported outcomes instrument with a 7-day recall period to measure AD disease control. Total score ranges from 0 to 24.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in ADCT score after 3, 6, 9, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  ADCT is a validated, brief and easy scored tool designed to evaluate patient-perceived control of atopic dermatitis, to foster communication between patients and their physicians and help appropriate decision-making. The ADCT is a 6-item patient-reported outcomes instrument with a 7-day recall period to measure AD disease control. Total score ranges from 0 to 24.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Recap of atopic eczema (RECAP) score after 3, 6, 9, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  Recap of atopic eczema (RECAP) is a seven-item questionnaire designed to capture the experience of eczema control in all ages and eczema severities. The RECAP can range from 0 to 28, where a lower score indicates a better outcome.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in RECAP score after 3, 6, 9, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  RECAP is a seven-item questionnaire designed to capture the experience of eczema control in all ages and eczema severities. The RECAP can range from 0 to 28, where a lower score indicates a better outcome.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Patient Oriented Eczema Measure (POEM) score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  POEM is a 7-item (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) questionnaire to assess frequency of disease symptoms with a scoring system of 0 to 28, the higher score indicating higher severity.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in POEM score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  POEM is a 7-item (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) questionnaire to assess frequency of disease symptoms with a scoring system of 0 to 28, the higher score indicating higher severity.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Dermatology Life Quality Index/Children's Dermatology Life Quality Index (DLQI/CDLQI) score after 6, 12, and 24 months of dupilumab therapy. | From baseline up to 24 months
  The Dermatology Quality of Life Index (DLQI) is a 10-item questionnaire to measure dermatology specific quality of life (QoL). The DLQI is designed for use in adults (patient's ≥ 16 years of age) and the CDLQI for patients < 16 years of age. Each question is scored on a four-point Likert scale.The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in Dermatology Life Quality Index (DLQI)/Children's Dermatology Life Quality Index (CDLQI) score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  The Dermatology Quality of Life Index (DLQI) is a 10-item questionnaire to measure dermatology specific quality of life (QoL). The DLQI is designed for use in adults (patient's ≥ 16 years of age) and the CDLQI for patients < 16 years of age. Each question is scored on a four-point Likert scale.The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Patient reported effectiveness and impact on QoL data: Mean Absolute Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance score after 6, 12, and 24 months of dupilumab therapy. | From baseline up to 24 months
  Patient-Reported Outcomes Measurement Information System® (PROMIS®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS® Sleep Disturbance Scale was developed to assess self-reported perceptions of sleep quality, sleep depth, and any perceived difficulties related to getting and staying asleep over a 7-day period. Response options for the sleep quality item range from: "Very poor (1)" to "Very good (5)" or from "Not at all (1)" to "Very much (5).
Patient reported effectiveness and impact on QoL data: Mean Percent Change from baseline in PROMIS sleep disturbance score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  Patient-Reported Outcomes Measurement Information System® (PROMIS®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. PROMIS® Sleep Disturbance Scale was developed to assess self-reported perceptions of sleep quality, sleep depth, and any perceived difficulties related to getting and staying asleep over a 7-day period. Response options for the sleep quality item range from: "Very poor (1)" to "Very good (5)" or from "Not at all (1)" to "Very much (5).
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in At baseline Questionnaire on Experience with Skin complaints (QES) score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  The Questionnaire on Experience with Skin Complaints (QES) [8] is a fully standardized self-rating instrument that focuses on the feelings of stigmatization of patients with different skin diseases and the coping with the stigma experience.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in At baseline Questionnaire on Experience with Skin complaints (QES) score after 6, 12, and 24 months of dupilumab therapy | From baseline up to 24 months
  The Questionnaire on Experience with Skin Complaints (QES) [8] is a fully standardized self-rating instrument that focuses on the feelings of stigmatization of patients with different skin diseases and the coping with the stigma experience.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Patient Global Assessment (PtGA) score after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The Global Patient Assessment is a 2-component questionnaire on symptom severity and the patient's overall satisfaction with their treatment.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in Patient Global Assessment (PtGA) score after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The Global Patient Assessment is a 2-component questionnaire on symptom severity and the patient's overall satisfaction with their treatment
Patient reported effectiveness and impact on QoL data: : Mean percent change from baseline in Asthma control questionnaire-5 (ACQ-5)-Scores, assessed only in patients with co-existing Asthma after 3, 6, 9,12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The ACQ-5 assesses asthma control using the 5-item ACQ-5 questionnaire.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Asthma control questionnaire-5 (ACQ-5)-Scores, assessed only in patients with co-existing Asthma) after 3, 6, 9,12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The ACQ-5 assesses asthma control using the 5-item ACQ-5 questionnaire.
Mean absolute change from baseline in Allergic Visual analogue Scales ([Allergic-VAS] only patients with co-existing overall allergic symptoms) after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  Patient reported effectiveness and impact on QoL data: will be assessed. Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Mean percent change from baseline in Allergic Visual Analogue Scales ([Allergic-VAS] only patients with co-existing overall allergic symptoms) after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From Baseline up to 24 months
  Patient reported effectiveness and impact on QoL data: will be assessed. Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in MACVIA-ARIA Sentinel Network Rhinitis Visual Analog Score (MASK-Rhinitis VAS score). | From baseline up to 24 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in MACVIA-ARIA Sentinel Network Rhinitis Visual Analog Score (MASK-Rhinitis VAS score) | From baseline up to 24 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in MACVIA-ARIA Sentinel Network conjunctivitis Visual Analog Score (MASK-conjunctivitis VAS score), after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy. | From baseline up to 24 months
  Only assessed in patients with co-existing allergic conjunctivitis. Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Mean percent change from baseline in MACVIA-ARIA Sentinel Network conjunctivitis Visual Analog Score (MASK-conjunctivitis VAS score) after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  Only assessed in patients with co-existing allergic conjunctivitis. Patient reported effectiveness and impact on QoL data: will be aVisual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. VAS is usually a horizontal 100 mm long scale with two opposing descriptors at its end points. The lower numbers indicate less severity, and the higher numbers indicate greater severity.
Patient reported effectiveness and impact on QoL data: Mean absolute change from baseline in Sinus Control Test (SCT) score, only assessed in patients with co-existing chronic rhinosinusitis after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The SCT involves four questions, three of which are answered using a 5-point Likert scale and one dichotomous question. The SCT total score is used to categorize patient control status into three groups: controlled (total score 0-3), partially controlled (total score 4-11), and uncontrolled (total score 12-16).
Patient reported effectiveness and impact on QoL data: Mean percent change from baseline in SCT score, only assessed in patients with co-existing chronic rhinosinusitis after 3, 6, 9, 12, 15, 18, and 24 months of dupilumab therapy | From baseline up to 24 months
  The SCT involves four questions, three of which are answered using a 5-point Likert scale and one dichotomous question. The SCT total score is used to categorize patient control status into three groups: controlled (total score 0-3), partially controlled (total score 4-11), and uncontrolled (total score 12-16).
Patient and treatment characteristics reported by the physician or patient: Socio -demographic data | At baseline
Patient and treatment characteristics reported by the physician or patient: Medical history of disease | At baseline
Patient and treatment characteristics reported by the physician or patient: Comorbidities/smoker status/alcohol usage | At baseline
Patient and treatment characteristics reported by the physician or patient: Prior systemic AD treatment (including balneophototherapy and/or UV therapy) | At baseline
Patient and treatment characteristics reported by the physician or patient: Current topical and/or systemic AD treatment of the last 4 weeks before baseline visit (dosage, type) | At baseline
Patient and treatment characteristics reported by the physician or patient: Current treatment for co-existing type 2 inflammatory and atopic diseases | At baseline
  Data reported for dosage and type of current treatment for co-existing type 2 inflammatory and atopic diseases.
Patient and treatment characteristics reported by the physician or patient: Reasons for initiating dupilumab treatment | At baseline
Patient and treatment characteristics reported by the physician or patient: Reasons for discontinuation of dupilumab treatment (if the discontinuation was before end of study) | Up to 24 months
  Reasons for discontinuation of dupilumab treatment (if the discontinuation was before end of study) will be collected at the discontinuation visit.
Patient and treatment characteristics reported by the physician or patient: Number of sick-leave days away from work/school due to AD | From baseline up to 24 months
Patient and treatment characteristics reported by the physician or patient: Number of medical appointments due to AD | From baseline up to 24 months
Patient and treatment characteristics reported by the physician or patient: Number of visits to alternative practitioners and complementary care physicians | From baseline upto 24 months
Patient and treatment characteristics reported by the physician or patient: Cost of non-reimbursable supplementary therapy [€/month] | From baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (55):
- Germany (55):
  - Investigational Site Number: 061, Aachen
  - Investigational Site Number: 092, Ahaus
  - Investigational Site Number: 066, Andernach
  - Investigational Site Number: 002, Berlin
  - Investigational Site Number: 003, Berlin
  - Investigational Site Number: 176, Berlin
  - Investigational Site Number: 077, Berlin
  - Investigational Site Number: 004, Berlin
  - Investigational Site Number: 174, Berlin
  - Investigational Site Number: 073, Berlin
  - Investigational Site Number: 059, Braunschweig
  - Investigational Site Number: 057, Buxtehude
  - Investigational Site Number: 028, Chemnitz
  - Investigational Site Number: 069, Cologne
  - Investigational Site Number: 072, Dresden
  - Investigational Site Number: 026, Dresden
  - Investigational Site Number: 032, Düren
  - Investigational Site Number: 043, Erlangen
  - Investigational Site Number: 064, Essen
  - Investigational Site Number: 184, Friedberg
  - Investigational Site Number: 055, Gera
  - Investigational Site Number: 007, Giessen
  - Investigational Site Number: 031, Gladbeck
  - Investigational Site Number: 078, Göttingen
  - Investigational Site Number: 087, Hamburg
  - Investigational Site Number: 088, Hamburg
  - Investigational Site Number: 020, Hamburg
  - Investigational Site Number: 086, Hamburg
  - Investigational Site Number: 169, Heidelberg
  - Investigational Site Number: 053, Heilbad Heiligenstadt
  - Investigational Site Number: 063, Jülich
  - Investigational Site Number: 186, Karlsruhe
  - Investigational Site Number: 016, Kiel
  - Investigational Site Number: 017, Kiel
  - Investigational Site Number: 183, Landsberg
  - Investigational Site Number: 038, Langenau
  - Investigational Site Number: 179, Leipzig
  - Investigational Site Number: 178, Mainz
  - Investigational Site Number: 185, Mainz
  - Investigational Site Number: 014, Mainz
  - Investigational Site Number: 013, Mannheim
  - Investigational Site Number: 018, Mölln
  - Investigational Site Number: 035, Mönchengladbach
  - Investigational Site Number: 050, München
  - Investigational Site Number: 076, Neubrandenburg
  - Investigational Site Number: 045, Nuremberg
  - Investigational Site Number: 042, Nuremberg
  - Investigational Site Number: 024, Oelde
  - Investigational Site Number: 082, Potsdam
  - Investigational Site Number: 172, Remscheid
  - Investigational Site Number: 177, Rostock
  - Investigational Site Number: 047, Wasserburg
  - Investigational Site Number: 019, Wismar
  - Investigational Site Number: 168, Wittlich
  - Investigational Site Number: 193, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org